CLINICAL TRIAL: NCT02171728
Title: A Phase I Open Label Dose Escalation Study of Continuous Once-daily Oral Treatment With BIBW 2992 in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation Study of Continuous Once-daily Oral Treatment With BIBW 2992 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.4
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental): dose escalation
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992

SUMMARY:
Investigation of maximum tolerated dose (MTD), safety, pharmacokinetics, pharmacodynamic parameters, and efficacy of BIBW 2992

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non-resectable and/or metastatic solid tumors, of types historically known to express EGFR and/or HER2 (Human Epidermal Growth Factor Receptor), who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment preferably patients with breast, colorectal or prostate cancer
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent that is consistent with International Conference on Harmonization - Good Clinical Practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2
* Patients recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies to CTC <=Grade 1
* Patients must be recovered from previous surgery

The 12 additional patients recruited at the MTD must also meet the following criteria:

* Measurable tumor deposits (RECIST) by one or more techniques (X-ray, CT, MRI) and/or recognized tumor markers such as prostate-specific antigen (PSA) (prostate cancer) or cancer antigen (CA) 125 (ovarian cancer)

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least eight (8) weeks, no history of cerebral edema or bleeding in the past eight (8) weeks and no requirement for steroids or anti-epileptic therapy
* Cardiac left ventricular function with resting ejection fraction CTC >=Grade 1
* Absolute neutrophil count (ANC) less than 1500/mm3
* Platelet count less than 100 000/mm3
* Bilirubin greater than 1.5 mg /dl (>26 μmol /L, SI unit equivalent)
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg/dl (>132 μmol/L, Système Internationale unit equivalent)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding Luteinizing Hormone-Releasing Hormone (LHRH) agonists, or other hormones taken for breast cancer, or bisphosphonates), or participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
* Treatment with an EGFR- or HER2 inhibiting drug within the past four weeks before start of therapy or concomitantly with this study (eight weeks for trastuzumab)
* Patients unable to comply with the protocol
* Active alcohol or drug abuse

A patient may be eligible for re-treatment after the previous course is finished. A patient will not be eligible if any of the following conditions are met:

* Patients with clinical signs of disease progression or if latest X-ray, CT or MRI reveals disease progression
* Cardiac left ventricular function CTC Grade ≥ 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria (except criterion 5) listed before as determined

  * On Day 28 of treatment period 1 or on Visit R1 of the current course when patient is entering the repeated treatment period (treatment period 2),
  * On Visit R5 of the previous course or on Visit R1/C1 of the current course when patient is in repeated treatment period (treatment courses 3 to 6) or when entering continuous treatment period (treatment course 7), or
  * On Visit C3 of the previous course or Visit C1 of the current course when patient is in continuous treatment period (treatment courses 8 to final discontinuation)
* Patient not recovered from any dose-limiting toxicity (DLT) 14 days after the last administration of BIBW 2992 in the previous course. Recovery is defined as return to baseline level or CTC Grade 1, whichever is higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-11; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of BIBW 2992 | up to 168 days
Incidence and intensity of Adverse Events according to Common Terminology Criteria (CTC version 3) | up to 23 months

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) for several time points | up to 28 days
Predose plasma concentration | Predose on day 8, 15, 22 and 27
Plasma concentration at 24 h following the first (C24,1) and the Day 27 dose (C24,27) | 24 hours after drug administration on day 24 and 27
Plasma concentration at 3 h following the first dose (C3,1) | 3 hours after the first dose on day 1
Maximum measured plasma concentration at steady state on Day 27 (Cmax,ss) | up to 24 hours after drug administration on day 27
Time from dosing to the maximum plasma concentration at steady state on Day 27 (tmax,ss) | up to 24 hours after drug administration on day 27
Terminal half-life at steady state (t1/2,ss) | up to 28 days
Mean residence time after oral administration at steady state (MRTpo,ss) | up to 28 days
Apparent clearance at steady state (CL/F,ss) | up to 28 days
Apparent volume of distribution during the terminal phase at steady state (Vz/F,ss) | up to 28 days
Objective tumor responses | up to 23 months
Correlation of EGFR (epidermal growth factor receptor), HER2, estrogen receptor (ER) and progesterone receptor (PrR) immunohistochemical status as based on tumor biopsies, or excisions obtained prior to this trial, with objective tumor responses | up to 23 months